CLINICAL TRIAL: NCT06018662
Title: Establishment of an Electronic Medication Management Application in a Pediatric Surgery Department
Brief Title: An Interventional Study to Establish a Medication Management Mobile Application for Pediatric Surgery Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mai Fawaz, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: A medication mobile app
Record Dates: First submitted 2023-08-03; First posted 2023-08-30 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Medication Management
Keywords: Pediatric surgery; Mobile application; Medication errors

STUDY DESIGN:
Intervention Model Description: Control group (138 patients): The medications selection and dosage will be performed according to the department policy without using the application.
  Intervention group (138 patients): The physicians use the application for appropriate medications selection and dosage calculation.
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Routine department therapy
- Interventional (Experimental): Anesthetics, antimicrobials and analgesics are selected and age/weight doses are calculated using the medication management mobile application
  Interventions: Other: A medication management mobile application

INTERVENTIONS:
Other: A medication management mobile application — A mobile application to select the most appropriate drugs for anesthetics, antimicrobials and analgesics, in addition to dose calculations
  Arms: Interventional

SUMMARY:
An interventional study that aims to design, establish and implement an electronic application for management of the usage of anesthetics, antimicrobials, and analgesics in a pediatric surgery department, and assess the impact of the implementation of an electronic medication management application on the appropriateness of medication use in a pediatric surgery department

DETAILED DESCRIPTION:
Mobile health (mHealth) refers to digital health technologies via mobile phones, tablets, and other electronic devices to enhance health outcomes. mHealth has started to have an impact on many health care and medical education aspects. With the increased number of smartphones and increasing interest in using mobile applications (apps), healthcare related mobile apps offer opportunities for advanced patient care allowing for better patient-provider communication. Within anesthesia, mobile apps were developed to play an important role; pre, intra- and postoperatively through providing patient-physician communication, reducing patient anxiety, and offering on-the-go education.

The development of medical mobile app is challenging. It incorporates producing an easy-to-use display with appropriate clinical information. Although many medication errors lead to little or no harm, some have overwhelming consequences for patients and, sometimes, for practitioners.

In pediatric patients, doses of anesthetics and other medications are calculated based on age and/or weight. Also, preparations often require further dilutions, specifically for younger patients like neonates and infants. These steps might increase risk for medication errors in pediatric anesthesia. For pediatric patients, it is important to use appropriate weight-based medication doses.

Anesthetics, Antimicrobials and Analgesics are the three drug classes that have shown the highest number of medication errors in the operating rooms of a pediatric surgery department. To provide an appropriate age and/or weight-based drug information, we will develop an electronic application to recommend the most appropriate drugs based on international guidelines and calculate doses for Anesthetics, Antimicrobials and Analgesics for pediatric patients in the operating rooms of a pediatric surgery department.

Aim of the study:

To design, establish and implement an electronic application for management of the usage of anesthetics, antimicrobials, and analgesics in a pediatric surgery department. To assess the impact of the implementation of an electronic medication management application on the appropriateness of medication use in a pediatric surgery department

Patients and methods:

Design:

Prospective, Interventional, Single-blinded, Randomized controlled study.

Setting:

The study will be conducted in the pediatric surgery department in the Children's hospital, Ain Shams University, Cairo, Egypt.

Patients:

Pediatric patients undergoing surgical operations.

Methods:

The study will be performed according to the following phases;

Phase 1: Application Design and Development

* The app will include all database required to provide appropriate medications and dosing for pediatric patients intraoperatively, postoperatively and on discharge.
* The user will need to enter the patient's age and weight, choose the type of surgery and the drug class and the app will show the appropriate medications and dosage.
* The app will present all the important information for drug administration by using; the British National Formulary for children (BNF-C) and Lexicomp online database as the dosage and administration references, and The American Health System Pharmacists (ASHP) clinical practice guidelines and UpToDate evidence-based clinical decision support resource will be used for to determine the appropriate anesthetics, antimicrobials, and analgesics for the surgeries to be included in the study.
* The researcher will ensure that the application will be displayed properly on the iPhone operating system (iOS) and Android mobile devices.

Phase 2: Simulation and Validation

* To test app validation, a simulation study will be conducted, where, data of patient's weight and age will be entered followed by selection of type of surgery and drug class.
* The app will provide the appropriate medications and dosage for each case scenario according to international treatment protocols and guidelines.
* Medications doses in each drug class will be calculated twice using the app and twice without the app, for each type of surgery.

Phase 3: Physicians' training Physicians will be trained on how to use the application for the selected types of surgeries. (List of surgeons will be accurately checked and randomly 50% of them will be allowed to enter training sessions for use of app in their practice (interventional group), while the rest 50% will not be given the training sessions in order to use the department policy (Control group).

Phase 4: Patients' recruitment and Application use in pre-, intra-, and post-operative stage Two hundred and seventy- six 276 patients will be randomly allocated to either control group or intervention group via simple randomization technique.

Control group (138 patients): The medications selection and dosage will be performed according to the department policy without using the app.

Intervention group (138 patients): The physicians use the app for appropriate medications selection and dosage calculation.

All patients will be followed up postoperatively during hospital stay. A follow-up form will be used to record all required data during hospitalization.

Cost estimation :

Estimated cost savings will be calculated based on reduction in medication errors by using the electronic app. This will include discontinuing unnecessary medications, modifications of dose or duration, no medication indication, and inappropriate medication combination.

Medication errors categories according to the National Coordinating Council for Medication Error Reporting and Prevention (NCC MERP) will be included in the cost saving analysis.

Phase 5: Usability testing An electronic form of the System Usability Scale (SUS), a widely used and validated 10-questions Likert scale, for measuring the app usability will be used to evaluate physicians' user experience of the app.

Phase 6: Follow-up All patients will be followed up for two weeks after discharge for any signs and symptoms of drug related problems or postoperative complications including pain, nausea, vomiting and surgical site infection using an electronic form or phone calls. A follow-up form will be used after discharge

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients undergoing any of the following surgeries: Circumcision, Inguinal Hernia, Hypospadias, Esophageal dilatation, uncomplicated Appendectomy, and complicated Appendectomy

Exclusion Criteria:

* Cardiac patients
* Diabetic patients
* Hypertensive patients
* Immunocompromised patients
* Patients with renal and/or liver failure

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 276 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Appropriateness of medications (anesthetics, antimicrobials, and analgesics) used in different types of surgeries | One year
  Determined through measuring incidence of medication errors and drug related problems

SECONDARY OUTCOMES:
Cost saving | One year
  Estimated cost savings will be calculated by calculating direct medical costs (including medication costs (multiplied by duration in days) of the intervened medications if the interventions belong to any of the mentioned types, laboratory tests, investigations and hospital care).
  Estimated cost avoidance will be calculated based on the probability score (probability of an adverse drug event in the absence of the intervention).
Cost avoidance | one year
  Estimated cost avoidance will calculated based on the probability of an adverse drug event in the absence of the mobile application
Time saving | one year
  Time saving resulting from using the application will be calculated in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Mai Fawaz, Master's degree, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No